CLINICAL TRIAL: NCT01336361
Title: Emerging Practice in Palliative Care: A Survey of the Perceptions of Physical Therapists Regarding the Role, Utilization, Goals, and Cultural Issues of Physical Therapy Intervention in the Palliative Care of Functionally Dependent Elderly.
Brief Title: Emerging Physical Therapy Practice in Palliative Care: A Survey of Perceptions of Physical Therapists
Status: Completed | Type: Observational
Sponsor: University of Montana (Other)
Responsible Party: Principal Investigator, Ellen Gakis-Day, Graduate Student, University of Montana
Other Study IDs: UMT IRB 52-11
Record Dates: First submitted 2011-04-13; First posted 2011-04-15 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Perception
Keywords: Palliative Care; Physical Therapy; Functionally Dependent Elderly
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Physical Therapists: Physical Therapists who are members of the American Physical Therapy Association (APTA) and live in the United States .
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — A one-time paper survey was mailed to subjects, along with a cover letter, explanation of the research study, and contact and informed consent information. A reminder postcard was sent to subjects approximately one week later, encouraging return of the completed survey.

SUMMARY:
The purpose of this study is to explore emerging physical therapy practice in palliative care, and the perceptions of physical therapists regarding their care of the functionally dependent elderly, including: (1) the role and utilization of palliative care intervention in current practice, (2) current and potential goal-setting practices which may relate to palliative care, and (3) therapists' awareness of cultural and psychosocial issues in patient care.

DETAILED DESCRIPTION:
Palliative Care is a growing medical practice specialty, however the level of physical therapist involvement and the particular roles for physical therapy in this evolving discipline are relatively unknown.

The purpose of this study was to explore emerging physical therapy practice in palliative care, and the perceptions of physical therapists regarding their care of the functionally dependent elderly, including the role and utilization of palliative care intervention in current practice, goal-setting practices which may relate to palliative care, and therapists' awareness of cultural and psychosocial issues in patient care.

ELIGIBILITY:
Inclusion Criteria:

* Physical Therapists who are members of the APTA and live in the United States
* Reported practice in an inpatient or home health setting

Exclusion Criteria:

None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Physical Therapists who are members of the APTA and live in the United States.
Sampling Method: Probability Sample
Enrollment: 228 (Actual)
Dates: Start 2011-04; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Perceptions of physical therapists regarding the role, utilization, goals, and cultural issues of physical therapy interventions in the palliative care of functionally dependent elderly. | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Ellen L Gakis-Day, BS PT, DPT, Principal Investigator — University of Montana
Locations (1):
- The Univeristy of Montana, Transitional Doctor of Physical Therapy Program, Missoula, Montana, United States